CLINICAL TRIAL: NCT03847194
Title: The Promoting Resilience in Stress Management (PRISM) Intervention: a Multisite Randomized Control Trial in Adolescents With Type 1 Diabetes
Brief Title: PRISM for Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joyce Yi-Frazier, Senior Clinical Research Scientist, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC-N130; R01DK121224 (NIH)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with 2 groups: PRISM (intervention) arm or standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISM Intervention Arm (Experimental): The goal of the intervention is to teach resilience resource skills for use in current or future stressful situations. The total intervention consists of two, 45-60 minute, one-on-one sessions approximately 2-4 weeks apart followed by a family meeting discussing the skills learned. Following the family session through week 12, participants receive bi-weekly "booster" contacts (1:1 check-in sessions with the interventionist) to practice/refresh skills and check-ins on how skills have been utilized. These boosters will then be delivered monthly in months 4-6. In addition, all PRISM participants have access to the digital PRISM app, which offers an interactive practice and tracking interface to continue enhancing skills.
  Interventions: Behavioral: Promoting Resilience in Stress Management (PRISM)
- Usual Care (No Intervention): Families in both randomization arms will receive usual medical care for diabetes, including psychosocial care provided by the mental health professionals affiliated with the diabetes clinic if needed. At both sites, every diabetes patient is cared for by a team of diabetes specialists which includes a provider (MD, Physician Assistant and/or Nurse Practitioner), dietician, and social worker. Subspecialty referrals for additional mental health or other support are made at the discretion of the primary diabetes provider.

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management (PRISM) — PRISM was developed based on stress and coping theory to be a brief, disease non-specific, skills-based intervention targeting adolescent resilience resources. PRISM teaches 4 pillars of resilience including stress management, goal setting, cognitive restructuring and benefit-finding in a one-on-one training program consisting of two, 45-60 minute sessions and supported by 6-months of booster sessions and a fully developed digital app for practice and tracking. A family session follows the individual sessions and was designed for the adolescent to communicate to his/her caregiver(s) the skills learned, and how the caregiver(s) could best support ongoing practice.
  Arms: PRISM Intervention Arm

SUMMARY:
It is well-known that adolescents with type 1 diabetes are at high risk for elevated diabetes-specific distress and poor glycemic control. This randomized controlled trial uses a novel, person-centered intervention designed to reduce diabetes distress and improve resilience skills, which the investigators hypothesize will in turn improve glycemic control and quality of life. If successful, results will greatly inform future research and clinical strategies aimed at improving outcomes among adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
Adolescents with type 1 diabetes (T1D) are at high risk for elevated diabetes distress, which greatly impacts their adherence, glycemic control (A1C), and overall quality of life (QOL). A potential barrier to improving these experiences may be that adolescents have few opportunities to develop the personal resources needed to handle adversity and manage stress. The "Promoting Resilience in Stress Management" (PRISM) intervention is a manualized, brief, skills-based intervention delivered in 2, 45-60 minute one-on-one sessions, followed by a family meeting and supplemented by booster sessions and a digital app. PRISM was developed from Stress and Coping theory and targets skills in stress-management and mindfulness, goal-setting, positive reframing, and meaning-making. All of these skills are associated with improved patient outcomes in diverse groups of adolescent populations with chronic/serious illness, and findings from a feasibility trial in adolescents with T1D showed PRISM to be highly feasible and desirable in this population. Further, a recent pilot randomized controlled trial among adolescents with cancer suggest PRISM is associated with improved perceptions of resilience, lower psychological distress, and higher QOL. This application proposes to build on our prior experience and fill three critical knowledge gaps: (1) PRISM's impact on A1C among adolescents with T1D; and (2) PRISM's impact on diabetes distress, self-reported adherence, and other patient-reported outcomes including resilience and QOL. This funding opportunity seeks to test interventions targeting diabetes distress for impact on glycemic control. Thus, the investigators propose a multi-site randomized controlled trial among N=160 adolescents (n=80 PRISM, n=80 Usual Care; ages 13-18) with the primary trial outcome of glycemic control 6-months post-enrollment. Time-in-range will be evaluated for participants on continuous glucose monitors as an exploratory aim. Secondary outcomes will include diabetes-distress, and patient-reported adherence, resilience, and quality of life. The investigators hypothesize PRISM will promote better glycemic control and improved diabetes distress than usual care. This application offers an opportunity to expand the body of knowledge regarding methodologically rigorous and evidence-based interventions for adolescents with T1D. Ultimately, this research has the potential to offer a practical, skills-based curriculum designed to improve outcomes for this high-risk group.

ELIGIBILITY:
Inclusion Criteria:

* • They are 13-18 years old

  * Diagnosed with T1D >12 months
  * Elevated distress score (PAID-T>=30)*****
  * Speak English fluently
  * Cognitively able to participate in intervention sessions and complete written surveys.

Exclusion Criteria:

* Patient refusal to participate (any age), or parental refusal to participate for patients less than 18 years of age

  * Cognitively or physically unable to participate
  * Patient unable to speak in the English language
  * Patient unable to read in the English or Spanish language
  * Adolescent is ward of state

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce P Yi-Frazier, PhD, Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
The DSMB, Lead RA and study team will regularly assess confidentiality of study participants. The following will be assessed and verified: All data will be maintained on secure computers in locked offices at Seattle Children's Research Institute (data collection center); the participant (and caregiver) has signed informed consent and HIPAA forms; all standard confidentiality/privacy rules and guidelines set by the Seattle Children's Research Institute are in compliance. A Certificate of Confidentiality will be obtained.

REFERENCES:
- [Derived] Yi-Frazier JP, Hilliard ME, O'Donnell MB, Zhou C, Ellisor BM, Garcia Perez S, Duran B, Rojas Y, Malik FS, DeSalvo DJ, Pihoker C, Bradford MC, Scott S, Devaraj S, Rosenberg AR. Promoting Resilience in Stress Management for Adolescents With Type 1 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2428287. doi: 10.1001/jamanetworkopen.2024.28287. PMID 39158914
- [Derived] O'Donnell MB, Scott SR, Ellisor BM, Cao VT, Zhou C, Bradford MC, Pihoker C, DeSalvo DJ, Malik FS, Hilliard ME, Rosenberg AR, Yi-Frazier JP. Protocol for the Promoting Resilience in Stress Management (PRISM) intervention: A multi-site randomized controlled trial for adolescents with type 1 diabetes. Contemp Clin Trials. 2023 Jan;124:107017. doi: 10.1016/j.cct.2022.107017. Epub 2022 Nov 21. PMID 36410689

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Otherwise eligible patients need to score 30 or above on the Problem Areas in Diabetes validated scale, indicating moderate distress.
Period: Overall Study
Arm/Group | PRISM Intervention Arm | Usual Care
Started | 85 | 87
Completed | 82 | 79
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: all consented and randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | PRISM Intervention Arm | Usual Care | Total
Number analyzed (Participants) | 85 | 87 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.6) | 15.7 (1.6) | 15.7 (1.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 35 | 33 | 68
  Female | 44 | 52 | 96
  Other | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 11 | 33
  Not Hispanic or Latino | 63 | 76 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 15 | 26
  White | 63 | 62 | 125
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 85 | 87 | 172
HbA1C [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.8 (1.9) | 8.6 (2.2) | 8.7 (2.1)
Insulin Pump use [Count of Participants; unit: Participants] | 55 | 60 | 115

OUTCOME MEASURES:

1. Primary Outcome: A1C
Description: hemoglobin A1C
Time Frame: 6 months
Population: intent to treat analysis
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | PRISM Intervention Arm | Usual Care
Number analyzed (Participants) | 85 | 87
percentage of glycosylated hemoglobin | 8.7 (1.8) | 8.6 (1.8)

2. Primary Outcome: Diabetes Distress
Description: Diabetes distress will be measured with the Problem Areas in Diabetes Scale, Teen Version. Higher scores indicate more distress. Total score ranges from 6 to 84.
Time Frame: 6 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM Intervention Arm | Usual Care
Number analyzed (Participants) | 85 | 87
score on a scale | 36.2 (12.5) | 39.9 (15.0)

3. Secondary Outcome: Resilience
Description: Resilience will be measured with the Connor-Davidson Resilience Scale. Higher scores indicate more resilience. Total score ranges from 0-40.
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM Intervention Arm | Usual Care
Number analyzed (Participants) | 85 | 87
score on a scale | 25.2 (6.8) | 25.7 (7.3)

4. Secondary Outcome: Diabetes-specific Quality of Life
Description: Diabetes-specific Quality of life will be measured using the adolescent self-report version of the Type 1 Diabetes and Life (T1DAL) which assesses diabetes-specific health-related quality of life (HRQOL) for people with type 1 diabetes (T1D). Higher scores indicate higher quality of life. Scale ranges 0-100, with higher scores indicating better quality of life.
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM Intervention Arm | Usual Care
Number analyzed (Participants) | 85 | 87
score on a scale | 56.9 (15.4) | 53.5 (15.0)

5. Secondary Outcome: Adherence
Description: Adherence will be measured with the Diabetes Self-Management Questionnaire (DSMQ). The DSMQ ranges from 0-35 with higher scores indicate higher adherence.
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRISM Intervention Arm | Usual Care
Number analyzed (Participants) | 87 | 85
score on a scale | 19.9 (7.0) | 17.9 (9.1)

ADVERSE EVENTS:
Time Frame: 12-months for each patient, between the period of January 2020 and November 2022.
Description: our definition of adverse event and/or serious adverse event does not differ from the clinical trials.gov definitions.
Arm/Group | PRISM Intervention Arm | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/85 | 1/87
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/87
Other Adverse Events (participants affected / at risk) | 0/85 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT03847194/Prot_SAP_000.pdf